CLINICAL TRIAL: NCT00490152
Title: Microbicide-Use Adherence, Acceptability, and Attitudes Among Sexually Active Young Women Participating in a Phase I Microbicide Trial (MTN 004) "Tell Juliana"
Brief Title: Microbicides Acceptability Among Sexually Active Young Women
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 062
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-05

CONDITIONS: HIV Infections
Keywords: HIV; Microbicide Gel; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — astodrimer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Participants use Vivagel™, applied vaginally twice daily for 14 days, and report their experiences via phone diary and teleconference.
  Interventions: Behavioral: Automated diary system
- 2: Participants use VivaGel™ Placebo, applied vaginally twice daily for 14 days, and report their experiences via phone diary and teleconference.
  Interventions: Behavioral: Automated diary system
- 3: Participants use HEC Placebo Gel (HEC Gel), applied vaginally twice daily for 14 days, and report their experiences via phone diary and teleconference.
  Interventions: Behavioral: Automated diary system

INTERVENTIONS:
Behavioral: Automated diary system — Participants will use a computerized phone diary to describe their experiences with the study product during the 14 days of the trial. They will have three teleconferences with "Juliana" to discuss the product and the technology used in the study. They will also have the opportunity to send emails to "Juliana" during the course of the study.
  Other Names: VivaGel™; 3% w/w SPL7013 Gel
  Groups: 1
Behavioral: Automated diary system — Participants will use a computerized phone diary to describe their experiences with the study product during the 14 days of the trial. They will have three teleconferences with "Juliana" to discuss the product and the technology used in the study. They will also have the opportunity to send emails to "Juliana" during the course of the study.
  Other Names: VivaGel™ Placebo
  Groups: 2
Behavioral: Automated diary system — Participants will use a computerized phone diary to describe their experiences with the study product during the 14 days of the trial. They will have three teleconferences with "Juliana" to discuss the product and the technology used in the study. They will also have the opportunity to send emails to "Juliana" during the course of the study.
  Other Names: HEC Placebo Gel; HEC Gel
  Groups: 3

SUMMARY:
ATN 062 is designed to gain scientific knowledge of microbicide-use adherence, acceptability, and attitudes among sexually active young women

DETAILED DESCRIPTION:
ATN 062 will take place in parallel to another study, MTN 004, "Phase I Study of the Safety and Acceptability of 3% w/w SPL7013 Gel (VivaGel™) Applied Vaginally in Sexually Active Young Women." ATN 062 will use quantitative and qualitative research methods. The quantitative method will consist of a computerized diary used by participants during the 14 days of the gel trial of MTN 004. The qualitative methods will include email messages sent by participants to a research assistant as a supplement to the diaries, as well as in-depth interviews through teleconferences to contextualize the recorded events. All study activities will be timed to coincide with those of MTN 004

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in MTN 004.
* Willing and able to provide written informed consent for ATN 062.
* Willing to participate as required by protocol, including completion of all assessments and follow-ups.

Exclusion Criteria:

* Refuses to have teleconferences audio recorded.
* Any social or medical condition that, in the investigator's opinion, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: HIV-negative women ages 18 to 24 years old who are non-pregnant, sexually active and enrolled in MTN 004 will be offered the option to enroll in ATN 062. Approximately half of the participants will be recruited in San Juan, PR, and the other half in Tampa, FL.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2007-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Microbicide use adherence as measured by a computerized phone diary | 21 days(through end of study)
Microbicide use adherence as measured by e-mail messages | 21 days (through end of study)
Microbicide use adherence as measured by in-depth interviews via teleconference | 21 days (through end of study)
Microbicide use acceptability as measured by a computerized phone diary | 21 days (through end of study)
Microbicide use acceptability as measured by e-mail messages | 21 days (through end of study)
Microbicide use acceptability as measured by in-depth interviews via teleconferences | 21 days (through end of study)
Microbicide use attitudes as measured by a computerized phone diary | 21 days (through end of study)
Microbicide use attitudes as measured by e-mail messages | 21 days (through end of study)
Microbicide use attitudes as measured by in-depth interviews via teleconferences | 21 days (through end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Carballo-Diéguez, PhD, Study Chair — HIV Center for Clinical and Behavioral Studies at the New York State Psychiatric Institute and Columbia University
Locations (3):
- United States (2):
  - University of South Florida College of Medicine, Tampa, Florida
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org